CLINICAL TRIAL: NCT02450032
Title: An Open, Multi-center Study to Determine the Antibody Response to 500µg G17DT Given at Weeks 0, 2, and 6 in the Treatment of Patients With Gastric Cancer
Brief Title: Study to Determine the Antibody Response to 500µg G17DT in Treatment of Patients With Gastric Cancer
Acronym: GC5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5
Record Dates: First submitted 2014-08-27; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- G17DT (Experimental): Treatment with 500µg/ 0.4mL dose of G17DT administered by intramuscular injection at 0, 2, and 6 weeks.
  Interventions: Biological: G17DT

INTERVENTIONS:
Biological: G17DT
  Other Names: Polyclonal Antibody Stimulator

SUMMARY:
This study was designed to investigate the antibody response generated by a 500µg dose of G17DT in patients with gastric cancer.

DETAILED DESCRIPTION:
Another study, GC2, initiated prior to the start of this study investigated the appropriate dose and dosing schedule for G17DT in patients with Stage I-III gastric cancer. The highest dose tested in the GC2 study was 250µg. This dose was well tolerated but was not considered sufficiently immunogenic. Since tolerability had not constrained dosing up to 250µg, the GC5 study was designed to investigate a 500µg dose administered as a regimen of 0, 2, and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed UICC Stage I, II or III gastric adenocarcinoma.
* Patients must have had a macroscopically curative resection for gastric cancer with absence of metastatic disease at the time of entry to the trial.
* Male or Female patients aged 18 years or older.
* Life expectancy of at least 3 months.
* WHO Performance Status of 0 to 1.
* Written informed consent

Exclusion Criteria:

* Gastric surgery within four weeks of baseline (Week 0, visit 2) or gastric surgery anticipated during the period of the study.
* History of other malignant disease within the previous five years, except nonmelanomatous skin cancer or in situ carcinoma of the uterine cervix.
* Previous use within the last four weeks, concomitant use of anticipated use in the period of study, of any anti-cancer therapies.
* Concomitant use of immunosuppressants, including systemic (i.e. oral or injected) corticosteroids.
* Females who were pregnant, planning to become pregnant or lactating.
* Patients taking part in another study involving an investigational or licensed drug or device in the three months preceding enrollment or during this study.
* Previous G17DT treatment.
* Haematologicial indicators:

Haemoglobin (Hb) < 10g/dL White blood cell count (WBC) < 4.0 x 10^9/L Platelets < 100 x 10^9/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-02; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Antibody Levels | Through Week 12
  Gastrin-17 antibodies are produced as a result of treatment with G17DT and the proportion of patients producing gastrin-17 antibodies was considered to be an appropriate measure of the immunogenicity of the dosing schedule under study.
Injection Site Reaction | Up to Week 12
  A physical examination for the presence of an abscess at the injection site was performed on each patient to assess tolerability to treatment at every posttreatment visit from Week 0 to Week 12.
Change in Subject's World Health Organization Performance Status | Through Week 12
  The subject's WHO performance status was evaluated at each visit up to Week 12 to assess changes in subject's ability complete normal daily activities.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization up to Week 24 or until death
  Vital status was monitored throughout the study. Patients were followed up to their death or the study completion date, 18 June 2001.
Adverse Events | Through week 12
  All adverse events reported during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stuart, MB ChB, Principal Investigator — Glasgow Royal Infirmary
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom